CLINICAL TRIAL: NCT06690060
Title: Mind Body Intervention for Chronic Migraine Headaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000778A
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Migraines; Chronic Pain
Keywords: Migraines; Headaches; Chronic Pain
MeSH Terms: conditions — Migraine Disorders; Chronic Pain; Headache

STUDY DESIGN:
Intervention Model Description: This is a cohort study in which all participants will receive the mind-body intervention. This is an exploratory study to help hone elements of the protocol through participant feedback and to determine variance and optimal survey measurement tools. We will not modify participant medication regimens and no pain or other medication prescriptions will be issued by the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-Body Intervention (Experimental): A Novel Mind body technique for the intervention will be taught in lectures and group discussion sessions
  Interventions: Behavioral: Mind-Body Intervention

INTERVENTIONS:
Behavioral: Mind-Body Intervention — The mind-body intervention will include regular 1 to 2 hour educational sessions and lectures, as well as supplemental reading material. In addition, individualized sessions will be offered each week for students who have additional questions and/or need additional time with the material.

SUMMARY:
The goal of this exploratory study is to test a mind-body interventional approach for the treatment of chronic migraines. The main goal is to obtain feasibility information on the protocol which has been used in other similar conditions. We will also evaluate multiple measurement tools in order to optimize a follow-up pilot study evaluating the impact of the protocol on migraines.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years of age)
2. Previously diagnosed with migraine headache based on ICHD-3 beta criteria 91
3. A score of ≥ 50 on the Headache Impact Test-6 self-report survey (moderate impact) 92
4. Presence of migraine headaches at least 5 days per month
5. Willing to engage in a Mind-Body intervention
6. Willing/able to participate in remote sessions

Exclusion Criteria:

1. Known history or suspicion of headaches due to organic cause (e.g. cancer, sinus infection, head trauma, cerebrovascular disease)
2. Diagnosis of other chronic pain syndromes that may cloud assessments (e.g. fibromyalgia, chronic idiopathic neck pain)
3. Diagnosis of cognitive impairment or dementia
4. Active addiction disorder, e.g. cocaine or IV heroin use, that would interfere with study participation
5. Major psychiatric comorbidity (e.g., schizophrenia). Anxiety and mild-moderate depression are not considered exclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
MIDAS | baseline, 4, 8, 13 and 20 weeks
  The 7-item Migraine Disability Assessment (MIDAS) is a commonly used and well validated self report survey for assessing migraine-related disability. Questions cover adverse life impacts (missed work, etc.), headache frequency, and headache intensity.
HIT-6 | baseline, 4, 8, 13 and 20 weeks
  The Headache Impact Test (HIT-6), a well-validated self reported survey, measures the impact of headaches on 6 aspects of health-related quality of life. A recent study has estimated that a change of 6-7 points was clinically meaningful in a cohort starting with a mean HIT-6 score of 65.0 (severe impact). The HIT-6 is a recommended NIH common data element for headache.

SECONDARY OUTCOMES:
Brief Pain Inventory Questionnaire (Short Form) | baseline, 4, 8, 13 and 20 weeks
  The Brief Pain Inventory questionnaire, which has been validated by Keller et al., will be utilized to gauge pain intensity during the duration of the study. The question about current pain medications will be modified slightly to include current frequency of use.
Pain Anxiety Symptom Scale (Short Form 20) | baseline, 4, 8, 13 and 20 weeks
  The short form Pain Anxiety Symptom Scale (PASS-20) is a 20 question survey assessing cognitive, avoidance, fear, and physiological anxiety due to pain. It has been validated by McCracken et al.
Somatic Symptoms Score (SSS-8) | baseline, 4, 8, 13 and 20 weeks
  The 8 question Somatic Symptoms Score (SSS-8) is a validated, abbreviated version of the 15 question Patient Health Questionnaire (PHQ)-15. SSS-8 survey questions pertain to pain, the gastrointestinal system, fatigue, and cardiovascular complaints.
Migraine Duration | baseline, 4, 8, 13 and 20 weeks
  We will ask participants to estimate how long, on the average, their migraine attacks lasted during the last two weeks.
NRS-11 | baseline, 4, 8, 13 and 20 weeks
  The 11-point Numeric Rating Scale (NRS-11) for headache pain intensity asks the patient to rate their pain intensity from 0 (no pain) to 10 (worst pain imaginable). The NRS-11 is recommended by the International Headache Society (IHS) for assessment of this parameter in clinical trials.
GAMS | baseline, 4, 8, 13 and 20 weeks
  The single question Global Assessment of Migraine Severity (GAMS) captures a patient's assessment of their overall disease severity. The GAMS is being tested at this stage because there is an abundance of published baseline and variance data for comparison.
Feedback on protocol | 13 weeks
  We will be receiving qualitative feedback on the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No